CLINICAL TRIAL: NCT05380323
Title: A Phase 1, Randomized, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability, and PK of LY3541105 Following Single Doses in Healthy/Overweight Participants and Multiple Doses in Overweight Participants
Brief Title: A Study of LY3541105 in Healthy and Overweight Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18350; J3S-MC-YEAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-05-01; First posted 2022-05-18 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Overweight; Healthy
Keywords: Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY3541105 (Part A) (Experimental): Single ascending doses of LY3541105 administered subcutaneously (SC).
  Interventions: Drug: LY3541105
- LY3541105 (Part B) (Experimental): Multiple ascending doses of LY3541105 administered SC.
  Interventions: Drug: LY3541105
- LY3541105 (Part C) (Experimental): Escalating doses of LY3541105 administered SC.
  Interventions: Drug: LY3541105
- Placebo (Part A) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo
- Placebo (Part B) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo
- Placebo (Part C) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3541105 — Administered SC.
  Arms: LY3541105 (Part A); LY3541105 (Part B); LY3541105 (Part C)
Drug: Placebo — Administered SC.
  Arms: Placebo (Part A); Placebo (Part B); Placebo (Part C)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3541105 in healthy and overweight participants. Blood tests will be performed to check how much LY3541105 gets into the bloodstream and how long it takes the body to eliminate it. The study will also evaluate the effects of LY3541105 on body weight and assess safety and tolerability of LY3541105. This is a 3-part study and may last up to 15, 26 and 24 weeks for each participant and may include up to 7, 15 and 16 visits in parts A, B and C, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation
* Male participants who agree to refrain from sperm donation and to use contraceptive methods and female participants not of childbearing potential
* Have a body mass index (BMI) in the range of greater than or equal to (>/=) 18.5 to less than (<) 32 kilogram per square meter (kg/m²), both inclusive (in Part A) or a BMI in the range of >/=27 to <40 kg/m², both inclusive (in Part B and C)
* Have had a stable weight for the last 3 months

Exclusion Criteria:

* Have history of diabetes (except gestational diabetes) or current diagnosis of diabetes
* Clinically significant abnormal electrocardiogram (ECG) at screening, as judged by the Investigator
* Have history or current evidence of a clinically significant cardiovascular condition

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Predose up to 26 weeks
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3541105 | Predose through day 43 (Part A) & day 78 (Part B)
  PK: AUC of LY3541105
PK: Time of Maximum observed Concentration (Tmax) of LY3541105 | Predose through day 43 (Part A) & day 78 (Part B)
  PK: Tmax of LY3541105
PK: Maximum Observed Concentration (Cmax) of LY3541105 | Predose through day 43 (Part A) & day 78 (Part B)
  PK: Cmax of LY3541105
Pharmacodynamics (PD): Absolute and Percentage Change from Baseline in Body Weight | Predose through week 26 (Part B Only)
  PD: Absolute and Percentage Change from Baseline in Body Weight

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - PRA International, Lenexa, Kansas
  - ICON Early Phase Services, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No